CLINICAL TRIAL: NCT06150001
Title: Reduction of Rocuronium-induced Injection Pain With Aspiration of Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202301309A3
Record Dates: First submitted 2023-11-15; First posted 2023-11-29 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia, General
Keywords: rocuronium; injection pain; withdrawal movement; rocuronium injection pain; rocuronium withdrawal movement
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dilute with normal saline (Placebo Comparator): Researchers will dilute rocuronium at a dose of 0.8mg/kg with 2mL of normal saline. The rocuronium mixture will be injected into participants intravenous catheter.
  Interventions: Drug: rocuronium-normal-saline mixture
- dilute with 2%lidocaine (Active Comparator): Researchers will dilute rocuronium at a dose of 0.8mg/kg with 2mL of 2%lidocaine. The rocuronium mixture will be injected into participants intravenous catheter.
  Interventions: Drug: rocuronium-lidocaine mixture
- dilute with investigator's blood (Experimental): Researchers will dilute rocuronium at a dose of 0.8mg/kg with 2mL of blood. The rocuronium mixture will be injected into participants intravenous catheter.
  Interventions: Drug: rocuronium-blood mixture

INTERVENTIONS:
Drug: rocuronium-normal-saline mixture — rocuronium will be pre-diluted with 2mL of normal saline. Researchers will inject the mixture into intravenous catheter.
  Other Names: rocuronium
  Arms: dilute with normal saline
Drug: rocuronium-lidocaine mixture — rocuronium will be pre-diluted with 2mL of 2%lidocaine. Researchers will inject the mixture into intravenous catheter.
  Other Names: rocuronium
  Arms: dilute with 2%lidocaine
Drug: rocuronium-blood mixture — Researchers will connect a syringe which contains 0.8mg/kg of rocuronium intravenous catheter, and then withdraw blood into the syringe. Finally inject the mixture into intravenous catheter.
  Other Names: rocuronium
  Arms: dilute with investigator's blood

SUMMARY:
The goal of this clinical trial is to learn about reduction of rocuronium injection pain in participants receiving general anesthesia. The main question aims to answer is whether diluting rocuronium with blood can reduce rocuronium injection pain. Rocuronium is a rapid onset muscle relaxant used in general anesthesia. Lidocaine is a local anesthetic. Researchers will

• inject diluted rocuronium in participant's intravenous catheter during induction. • record withdrawal movement and rocuronium onset time and duration measured by train-of-four (TOF).

Researchers will compare between rocuronium diluted with blood, lidocaine and normal saline to see if blood can reduce rocuronium injection pain.

DETAILED DESCRIPTION:
This clinical trial uses a random table for sequential randomization, randomly assigning subjects to 3 groups, each consisting of 40 participants.

Researcher will confirm the patency of peripheral intravenous lines before induction. If peripheral intravenous lines cannot be used, they will be readministered at another injection site. If there are difficulties in peripheral intravenous injection, the participant will need to withdraw from this clinical trial. The neuromuscular monitoring device (NMT) is installed before the start of the clinical trial to monitor the effects of the drug. To avoid influencing the final results, fentanyl and 2%lidocaine will not be administered before injecting rocuronium. Anesthesia induction begins with the administration of oxygen through a mask to assist breathing. Initially, propofol is injected at a dose of 1.5 to 2mg/kg. Once the participant is confirmed to have lost consciousness, researchers will inject diluted rocuronium immediately, with an injection speed of 10 to 15 seconds. The dose of rocuronium for each participant is 0.8 mg/kg. The first group is pre-diluted with 2mL of normal saline, the second group with 2mL of 2%lidocaine, and the third group with 2mL of the participant's blood. To avoid clotting of blood, the procedure of the third group involves using a syringe containing rocuronium to withdraw 2mL of blood from the vein, followed by simultaneous injection into the intravenous line. The NMT is used to monitor the drug's effects, defining the onset time as the time from rocuronium injection to the disappearance of train-of-four (TOF) count T1 and the duration of action as the time from rocuronium injection to the appearance of TOF count T1.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the written informed consent form.
* Males and females aged 18 to 65.
* Undergoing endotracheal intubation under general anesthesia.
* Anesthesia physical status classification II or below.

Exclusion Criteria:

* estimated glomerular filtration rate less than 60
* History of cirrhosis or liver failure
* Neuromuscular disease or neurological symptoms
* Mental illness
* Arrhythmia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
withdrawal movement by 4-point-scale | From enrollment to the end of assessment at thirty minutes.
  withdrawal movement is measured by 4-point-scale. Zero is equivalent to no withdrawal movement. One is equivalent to withdrawal movement involving wrist joint. Two is equivalent to withdrawal movement involving elbow joint. Three is equivalent to withdrawal movement involving shoulder joint

SECONDARY OUTCOMES:
onset time | From enrollment to the end of assessment at 3 minutes.
  onset time is defined by injection of rocuronium mixture to the disappearance of Train-of-four count T1.
duration of action | From enrollment to the end of assessment at one hour.
  Duration of action is defined by injection of rocuronium mixture to appearance of Train-of-four count T1.

CONTACTS AND LOCATIONS:
Locations (1):
- ChangGung MH, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No